CLINICAL TRIAL: NCT03408366
Title: Feasibility of Assessing Wound Perfusion at the Time of Laparotomy Closure
Brief Title: A Study Assessing Circulation Around Surgical Incisions at the Time of Laparotomy Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-650
Record Dates: First submitted 2018-01-17; First posted 2018-01-24 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Laparotomy
Keywords: Laparotomy; Surgical Incisions; Wound Perfusion; 17-650
MeSH Terms: conditions — Surgical Wound | interventions — Laparotomy

STUDY DESIGN:
Intervention Model Description: Twenty consecutive patients will be enrolled: the first 10 will have skin closure with staples, and the second 10 will have skin closure with a running subcuticular suture.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women having a Laparotomy (Experimental): The first 10 patients enrolled will undergo skin closure with staples. The next 10 patients enrolled will undergo skin closure with a running subcuticular suture.to evaluate skin perfusion using the Spectrum NIR imaging system following intravenous injection of ICG in all patients. Patients will be assigned skin closure with either running subcuticular suture or skin staples in a sequential, nonrandomized fashion before the procedure. After the planned surgical procedure is complete, ICG will be injected intravenously. Video of the incision will be recorded. After skin closure is complete, a second intravenous bolus of ICG (same dose as previously injected) will be given. Video of the incision will again be recorded. Measurement of perfusion will subsequently be performed by video analysis at the previously described three predefined points along the incision after surgery is complete and again after skin closure.
  Interventions: Procedure: Laparotomy; Other: ICG; Other: Spectrum NIR imaging system

INTERVENTIONS:
Procedure: Laparotomy — Laparotomy via vertical midline incision and after the planned surgical procedure is complete.
Other: ICG — ICG will be injected intravenously ICG is a fluorescent iodide dye.
Other: Spectrum NIR imaging system — The Spectrum NIR imaging system uses a handheld camera that emits light in the NIR range.

SUMMARY:
This study is being done to find out if Spectrum Near-Infrared (NIR) imaging with Indocyanine Green (ICG) dye can help measure blood flow around an incision before and after the surgeon closes the incision with staples or sutures.

The Spectrum NIR imaging system uses a handheld camera that produces a special type of light that can help surgeons see things during surgery that are difficult to see with the naked eye, for example, cancer tissue versus healthy tissue. Spectrum NIR imaging has been approved by the Food and Drug Administration (FDA) as a tool that is widely used during surgery.

ICG dye is a sterile solution that can be seen with Spectrum NIR imaging. This dye, used with Spectrum NIR imaging, allows surgeons to see blood flow to parts of the body during and after surgery. Making sure that there is enough blood flow to the surgical site helps to promote a less complicated recovery.

ELIGIBILITY:
Criteria for Eligibility Prior to Surgery

Inclusion Criteria:

* Woman undergoing a laparotomy procedure via a vertical midline incision for any indication with the Gynecology Service at MSK
* Age ≥18 years

Exclusion Criteria:

* Women with hepatic dysfunction as evidenced by elevated transaminases
* Women with a history of cirrhosis or other chronic liver disease
* Women with an allergy to iodine
* Women undergoing laparoscopic or minimally invasive surgery

Criteria for Eligibility Post-Surgery

Inclusion Criteria:

* Woman undergoing a laparotomy procedure via a vertical midline incision for any indication with the Gynecology Service at MSK
* Age ≥18 years

Subject Exclusion Criteria:

* Women with laparotomy incisions unable to be closed primarily due to tissue or fascial damage
* Women with transverse laparotomy incisions
* Women with laparotomy incisions left open due to a case classification as "contaminated" or "dirty"

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman undergoing a laparotomy procedure
Enrollment: 20 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
percentage of cases with successful perfusion measurements | 1 year
  Feasibility will be determined by the percentage of cases with successful perfusion measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Abu-Rustum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memoral Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre (Consent only), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm